CLINICAL TRIAL: NCT04797754
Title: Systematic Development and Test-Retest Reliability of Electronic Instrumental Activities of Daily Living Satisfaction Assessment (EISA)
Brief Title: Systematic Development and Test-Retest Reliability of EISA
Acronym: EISA
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Abbas Quamar, Graduate Student Researcher, University of Pittsburgh
Other Study IDs: PRO17030604
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Disabilities Physical; Sensory Disorder
Keywords: Assistive Technology; Activities of Daily Living; Information & Communication Technology; Outcome Assessment
MeSH Terms: conditions — Sensation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this proposed study, is the development and validation of EISA, a Self-report outcome measurement tool, for assessing the satisfaction of everyday functional needs, for consumers using Electronic Assistive Devices (EADs) as the primary means to complete Instrumental Activities of Daily Living (IADLs). The EISA outcome measure is proposed to be designed as a questionnaire that can be self or interview-administered to users of EADs. The development of EISA shall be modeled along the lines of development of the self-report outcome measure, Functional Mobility Assessment (FMA) (Kumar et al., 2013). The proposed tool EISA, would serve as a dynamic gage, for assessing perceived user function, related to using EADs for completing IADLs. The instrument is proposed to undergo systematic development in three phases. In phase 1, an initial pool of potential EISA items shall be generated, based on literature review data.

In phase 2, content experts (clinician and EADs user) review panels, shall assess the initial pool of potential EISA items for further content validity. The objective of phase 3, would be a validation of the first iteration of EISA, by establishing reliability for test-retest administration and internal consistency, at acceptable levels, by 25-100 EADs users. Statistical analysis for test-retest reliability and internal consistency estimation shall be carried out in phase 3 of the study, using Statistical Package for the Social Sciences (SPSS) version 24 software.

DETAILED DESCRIPTION:
Objective: The purpose of this proposed study, is the development and validation of EISA, a Self-report outcome measurement tool, for assessing satisfaction of everyday functional needs, for consumers using EADs as the primary means to complete IADLs. The EISA outcome measure is proposed to be designed as a questionnaire that can be self or interview administered to users of EADs. Development of EISA shall be modeled along the lines of development of the self-report outcome measure, FMA (Kumar et al., 2013). The proposed tool EISA would serve as a dynamic gauge, for assessing perceived user function, related to using EADs for completing IADLs.

Specific Aims:

The instrument is proposed to undergo systematic development in three phases. In Phase 1, an initial pool of potential EISA items shall be generated, based on literature review data.

In Phase 2, content experts (clinician and EADs user) review panels, shall assess the initial pool of potential EISA items for further content validity. The objective of phase 3, would be validation of the first iteration of EISA, by establishing reliability for test-retest administration and internal consistency, at acceptable levels, by 25-100 EADs users.

Statistical analysis for test-retest reliability and internal consistency estimation shall be carried out using Statistical Package for the Social Sciences (SPSS) version 24 software, in Phase 3 of the study.

Background: Briefly describe previous findings or observations that provide the background leading to this proposal. It cannot be stressed enough, that for both able-bodied individuals and PWD, having access to ICT, is no longer a luxury, but rather, a basic necessity, to cope with the current technology based lifestyle. Furthermore, having equal and timely access to IT for PWD is imperative to enable them to live independently and have a high Quality of Life. Moreover, this equal and timely access not only provides increased life options for PWD but also, wider economic benefits for the society at large. However, currently, several factors are impeding this equal and timely access to ICT for PWD. These factors include (1) lack of an outcome measure specifically designed and validated to assess the satisfaction of everyday functional needs related to EAD; (2) inappropriateness, impracticality, apart from lack of clinical utility and psychometric validation of existing outcome measures to assess the satisfaction of everyday functional needs of PWD, related to EADs; (3) continual and fast-paced, disruptive innovations very often rendering essential services inaccessible for PWD. Therefore, to fill this unmet need, as well as, to enable PWD to have equal opportunity with able-bodied individuals to tap their optimal potential, this study proposes the development and validation of a self-report outcome measure, EISA, specifically designed to assess satisfaction of everyday functional needs of PWD, related to EADs.

Significance: In this day and age of IT, it is crucial for PWD to have access to EAD that matches their individualized needs and enables them to achieve their optimal potential. Nevertheless, as can be gleaned from the aforementioned analysis, currently there is no good outcome tool for the assessment of user-satisfaction in performing functional needs with EADs.

ELIGIBILITY:
Inclusion Criteria:

1. Should be an existing user of EADs for at least 3 months
2. Must be 18 years of age or older
3. Should be capable of cognitively reading instructions and answering questions within the Qualtrics online research platform

Exclusion Criteria:

1. Unable to read English
2. Unable to independently answer or have assistance from someone to answer the survey questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for the proposed EISA outcome measure would be Persons with Disabilities (PWD) who use EADs as their primary means for completing IADLs. Recruitment of EADs users shall be carried out in a targeted manner, through an invitation to participate in the study, by clinicians at (1) University of Pittsburgh Medical Center (UPMC) Center for Assistive Technology (CAT); (2) Hiram G. Andrews Center (HGAC) Center for Assistive and Rehabilitative Technology (CART); (3) The Ohio State University (OSU) Assistive Technology Clinic; and (4) the Veterans Administration Assistive Technology Labs.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Electronic Instrumental activities of daily living Satisfaction Assessment (EISA) | 6 months
  The EISA is a self-report outcome measurement tool, for assessing satisfaction of everyday functional needs, for consumers using Electronic Assistive Devices (EADs) as the primary means to complete IADLs. The EISA outcome measure is proposed to be designed as a questionnaire that can be self or interview administered to users of EADs.

OTHER OUTCOMES:
Demographic Questionnaires | Six Months
  This questionnaire is used to collect demographic information about the study cohort including age, experience using internet-connected EADs, level of education completed, if disabled, type of disability, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Schmeler, PhD, Study Director — University of Pittsburgh, School of Health and Rehabilitation Professionals
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The data will be uploaded by study participants to the Qualtrics Research Platform that is secure, encrypted and password protected. Only study personnel will have access to download unidentified data on excel sheets for data analysis.

REFERENCES:
- [Background] Donnelly C, Carswell A. Individualized outcome measures: a review of the literature. Can J Occup Ther. 2002 Apr;69(2):84-94. doi: 10.1177/000841740206900204. PMID 11977872
- [Background] Kumar A, Schmeler MR, Karmarkar AM, Collins DM, Cooper R, Cooper RA, Shin H, Holm MB. Test-retest reliability of the functional mobility assessment (FMA): a pilot study. Disabil Rehabil Assist Technol. 2013 May;8(3):213-9. doi: 10.3109/17483107.2012.688240. Epub 2012 May 22. PMID 22612721
- [Background] Scherer M, Jutai J, Fuhrer M, Demers L, Deruyter F. A framework for modelling the selection of assistive technology devices (ATDs). Disabil Rehabil Assist Technol. 2007 Jan;2(1):1-8. doi: 10.1080/17483100600845414. PMID 19263548
- [Background] Schmitter-Edgecombe M, Parsey C, Lamb R. Development and psychometric properties of the instrumental activities of daily living: compensation scale. Arch Clin Neuropsychol. 2014 Dec;29(8):776-92. doi: 10.1093/arclin/acu053. Epub 2014 Oct 25. PMID 25344901
- [Background] Demers L, Monette M, Descent M, Jutai J, Wolfson C. The Psychosocial Impact of Assistive Devices Scale (PIADS): translation and preliminary psychometric evaluation of a Canadian-French version. Qual Life Res. 2002 Sep;11(6):583-92. doi: 10.1023/a:1016397412708. PMID 12206579
- [Background] Day H, Jutai J, Campbell KA. Development of a scale to measure the psychosocial impact of assistive devices: lessons learned and the road ahead. Disabil Rehabil. 2002 Jan 10-Feb 15;24(1-3):31-7. doi: 10.1080/09638280110066343. PMID 11827152